CLINICAL TRIAL: NCT00218556
Title: Preventing Depression in MMT Patients on Interferon
Brief Title: Preventing Depression in Methadone Maintenance Patients Receiving Hepatitis C Treatment - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Associate Professor (Research), Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIDA-16797-1; R01-16797-1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2015-10

CONDITIONS: Depressive Disorder, Major; Hepatitis C
Keywords: Hepatitis C, Depressive Symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Hepatitis C; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Depression prevention (Experimental): Cognitive behavioral treatment for depression.
  Interventions: Behavioral: Cognitive behavioral treatment for depression
- Control (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: Cognitive behavioral treatment for depression — Cognitive behavioral intervention to prevent depressive symptoms during treatment for hepatitis C
  Arms: Depression prevention

SUMMARY:
The purpose of this study is develop and test a cognitive-behavioral intervention to prevent depression in methadone maintenance patients receiving medical treatment for hepatitis C.

DETAILED DESCRIPTION:
The purpose of this study is to develop a CBT-D intervention tailored to meet the needs of MMT patients undergoing antiviral treatment for hepatitis C. In the first phase of this project (Year 1), we will develop and pilot the intervention with 20 patients. In the second phase of the project (Years 2 and 3), we will conduct a preliminary, randomized trial with 60 MMT patients to examine the efficacy of the CBT-D intervention relative to standard care condition (SC).

We expect that, relative to the SC condition, participants randomized to the CBT-D condition will have decreased likelihood of depression-related antiviral treatment failure, will report lower levels of depressive symptoms, will complete more IFN injections, will have lower HCV RNA levels, and will have fewer illicit drug use days. If the efficacy of this intervention can be established in this trial and in subsequent clinical trials, MMT patients who elect to undergo antiviral therapy will have a valuable adjunct or alternative to the use of antidepressants to prevent depression. If found to be efficacious, this intervention will maximize the receipt of IFN treatment by MMT patients, thereby aiding in the prevention of liver failure, hepatocellular carcinoma, and liver-related death among those with HCV.

ELIGIBILITY:
Inclusion Criteria:

* Currently undergoing HCV treatment at RIH
* Enrolled in MMT for at least 6 months

Exclusion Criteria:

* Current major depressive episode
* Current suicidality
* Currently taking antidepressant medication
* Received HCV treatment in past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
depression-related antiviral treatment failure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Ramsey, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States